CLINICAL TRIAL: NCT05068895
Title: Assessment of Metabolic Profiles of Lower Extremity Arterial Disease in Patiens Withe Type 2 Diabetes Via LC-MS-based Nontargeted Metabolomic Approach
Brief Title: Assessment of Metabolic Profiles of Lower Extremity Arterial Disease in Patiens Withe Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: MP of LEAD
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Angiopathies; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Lower extremity artery disease; Metabolic Profiles; Metabolic biomarkers; Metabolomics; iquid chromatography-mass spectrometry
MeSH Terms: conditions — Diabetic Angiopathies; Diabetes Mellitus, Type 2 | interventions — Liquid Chromatography-Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group1: Volunteers with normal glucose tolerance.
  Interventions: Other: liquid chromatography-mass spectrometry
- Group2: type 2 diabetic patients without microvascular (retinopathy, nephropathy or neuropathy) or macrovascular (coronary, cerebrovascular or lower extremity arterial disease) complications.
  Interventions: Other: liquid chromatography-mass spectrometry
- Group3: type 2 diabetic patients with lower extremity artery disease diagnosed through the measurement of ABI (the ratio of ankle-to-brachial systolic blood pressure).
  Interventions: Other: liquid chromatography-mass spectrometry

INTERVENTIONS:
Other: liquid chromatography-mass spectrometry — Metabolomics is a rapidly evolving high-throughput technology that allows the measurement of the entire complement of metabolites generated by biochemical reactions under certain conditions in biological fluids or tissues. This technology has been used extensively to identify biomarkers in various cancers, nervous system diseases, cardiovascular diseases, pituitary diseases, and other diseases. The identification of biomarkers can be clinically useful for a more accurate diagnosis, prognosis, and treatment choice as well as disease monitoring. Among mass spectrometry (MS) methods, liquid chromatography-mass spectrometry (LC-MS) has been recognized as a robust metabolomics tool and has been widely applied in metabolite identification and quantification due to its high sensitivity, peak resolution, and repro- ducibility.
  Other Names: Metabolomics

SUMMARY:
The prevalence of lower extremity arterial disease (LEAD) in patients with diabetes increases significantly and are characterized with obvious arteriosclerosis that are caused by multiple metabolic disorders. Metabolomics measures the metabolites in biological fluids or tissues that generated under certain conditions via rapidly evolving high-throughput technology. Herein, the investigators designed the study to characterize the serum metabolic profiles of LEAD patients and identify metabolic biomarkers using metabolomics. The serum of volunteers, type 2 diabetes mellitus(T2DM) patients with or without LEAD were collected and analyzed using liquid chromatography-mass spectrometry(LC-MS) coupled with a series of multivariate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 18 to 100 years old
* Signed informed consent and agreed to participate in this study
* The diagnosis of T2DM is based on standard criteria recommended by WHO since 1999
* The diagnosis of T2DM patient with LEAD is based on standard criteria recommended by Chinese guideline on prevention and management of diabetic foot (2019 edition)(II).

Exclusion Criteria:

* younger than 18 years old or older than 100 years old
* acute infection during the preceding 3 months
* drugs or alcohol addicts
* cancer
* type 1 diabetes
* patients with mental abnormality who are uncooperative with this study
* pregnant or lactating women
* refuse to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We collected serum samples and clinical data of 74 volunteers and patients with T2DM who hospitalized in our department from June 2021 to September 2021.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-09 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Metabolic profiles of lower extremity artery disease | 4 months
  LC-MS analysis will be performed using a Q ExactiveTM HF-X liqiud chromatograph system coupled with a Thermo ScientificTM OrbitrapTM mass spectrometer according to a previously published procedure to detect the peak, identify the metabolites and perform the PCA and OPLS-DA analyses to better visualize the subtle similarities and differences among the complex datasets.

SECONDARY OUTCOMES:
Potential biomarker analysis for discrimination | 4 months
  Screening for potential biomarkers will be performed according to the VIP value (VIP > 1.0) and significance test (P < 0.05) from the OPLS-DA model.
Pathway analysis of differential metabolites | 4 months
  Conducting pathway analysis for the significant metabolites identified by using MetaboAnalyst.

CONTACTS AND LOCATIONS:
Overall Officials: Zhencheng Yan, MD, Study Director — The third hospital affiliated to the Third Military Medical University
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] You M, Liu Y, Wang B, Li L, Zhang H, He H, Zhou Q, Cao T, Wang L, Zhao Z, Zhu Z, Gao P, Yan Z. Asprosin induces vascular endothelial-to-mesenchymal transition in diabetic lower extremity peripheral artery disease. Cardiovasc Diabetol. 2022 Feb 15;21(1):25. doi: 10.1186/s12933-022-01457-0. PMID 35168605